CLINICAL TRIAL: NCT05422742
Title: Influence of Scaling and Root Planing With Minocycline Microspheres on the Composition and Functional Characteristics of Subgingival Microbiome Communities
Brief Title: Influence of SRP With MM on the Composition and Functional Characteristics of Subgingival Microbiome Communities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008078967
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SRP (Active Comparator): Scaling and rooting planning
  Interventions: Procedure: Scaling and Root Planing (SRP)
- SRP + MM (Experimental): Scaling and rooting planning in combination with minocycline microspheres
  Interventions: Procedure: SRP + MM
- Periodontally-Healthy Subjects (No Intervention): No Intervention

INTERVENTIONS:
Procedure: SRP + MM — Subjects will be randomized into either SRP only or SRP +MM. Periodontal therapy will consist of one visit full-month SRP alone or in-combination with MM placed at all sites regardless of probing pocket depth. Each site will recieve 1mg of MM for a total of 6mg of MM per tooth.
  Arms: SRP + MM
Procedure: Scaling and Root Planing (SRP) — Procedure involving removal of dental plaque and calculus (scaling or debridement) and then smoothing, or planing, of the (exposed) surfaces of the roots, removing cementum or dentine that is impregnated with calculus, toxins, or microorganisms, the etiologic agents that cause inflammation.
  Arms: SRP

SUMMARY:
The purpose of this study is to characterize the effect of minocycline microspheres (MM) administered as an adjunct to scaling and rooting planning (SRP) on the subgingival community composition and metatranscriptome functional profile, in comparison to a group treated with SRP only and to periodontally-healthy subjects.

DETAILED DESCRIPTION:
Patients attending the West Virginia University School of Dentistry Clinics will be invited to participate in this study. Thirty periodontitis patients (stage II, III or IV) with ≥4 teeth with a probing pocket depth (PPD) >4 mm; at least 1 tooth with a PPD >6 mm and clinical attachment loss (CAL) ≥2 mm, and radiographic evidence of bone loss will be recruited.

Clinical examination will include measurement of clinical attachment loss (CAL), probing pocket depth (PPD), bleeding on probing (BOP), and plaque score (PS) at 6 sites per tooth. Furcation involvement (FI) will also be recorded. Radiographic examination will include full-mouth radiographic series. Patients will receive a clinical examination at baseline (V1, before periodontal therapy), and their subgingival plaque biofilms will be sampled at a second visit (V2) two weeks after this initial exam to collect subgingival plaque not disrupted by the examination procedures.

Subjects will be then randomized to one of two groups: SRP only and SRP + MM. Periodontal therapy will consist of one visit (V3) full-mouth SRP alone or in combination with MM placed at all sites regardless of PPD. Each site will receive 1mg of MM for a total of 6mg of MM per tooth. In this manner we will also evaluate whether MM modifies the microbiome of shallow sites, since subgingival microbiome dysbiosis affects shallow sites of subjects with periodontitis and therefore represents a risk for future disease progression.

Subjects will be evaluated 2 months after receiving periodontal therapy (V4). At this visit subgingival plaque samples will be collected and clinical outcomes evaluated. Clinical examinations and plaque collection will be conducted by one calibrated examiner.

Fifteen periodontally-healthy subjects will also be recruited from the West Virginia University School of Dentistry Clinics. Subjects will receive a clinical examination and their subgingival communities sampled at the same visit (V1).

ELIGIBILITY:
Inclusion Criteria for randomized participants:

* Have at least 20 natural teeth with a diagnosis of Periodontitis (stage II, III, or IV).

Inclusion Criteria for periodontally-healthy participants:

* Diagnosis of healthy periodontium defined as ≤9% of sites bleeding on probing with absence of interproximal attachment loss and bone loss

Exclusion Criteria for all participants:

* Pregnancy or lactation
* Patients with diabetes mellitus or any other systemic disease that can modify periodontitis
* Current smokers
* Current use of f any medication with known effects on periodontitis
* Use of non-steroidal anti-inflammatory drugs
* Use of local or systemic antibiotics within the last 3 months
* Subjects with conditions requiring prophylactic antibiotics
* Subjects allergic to any of the tetracyclines
* Professional dental cleaning within the last 3 months
* SRP or surgical periodontal therapy in the previous year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Attachment Loss (SRP + MM) | baseline to 2 months post procedure
  Change in Clinical Attachment Loss which is a routine clinical measure of periodontal health (measured in mm) from baseline to 2 months post procedure
Change in Clinical Attachment Loss (SRP only) | baseline to 2 months post procedure
  Change in Clinical Attachment Loss which is a routine clinical measure of periodontal health (measured in mm) from baseline to 2 months post procedure
Probing Pocket Depth (SRP + MM) | Baseline to 2 months post procedure
  Change in Probing depth is a routine clinical measure of periodontal health (measured in mm)
Probing Pocket Depth (SRP only) | Baseline to 2 months post procedure
  Change in Probing depth is a routine clinical measure of periodontal health (measured in mm)
Bleeding on Probing (SRP + MM) | Baseline to 2 months post procedure
  Change in Bleeding on Probing is a measure of inflammation and determined as the percent of bleeding sites that are measured at 6 sites per tooth
Bleeding on Probing (SRP only) | Baseline to 2 months post procedure
  Change in Bleeding on Probing is a measure of inflammation and determined as the percent of bleeding sites that are measured at 6 sites per tooth
Plaque Score (SRP + MM) | Baseline to 2 months post procedure
  Change in O'Leary plaque score. Plaque score will be assessed dichotomously. Score 1 when plaque is identifiable using a dental probe or score 0 when no plaque is present. Following this assessment, plaque score is calculated by dividing the number of plaque containing surfaces by the total number of surfaces examined.
Plaque Score (SRP only) | Baseline to 2 months post procedure
  Change in O'Leary plaque score. Plaque score will be assessed dichotomously. Score 1 when plaque is identifiable using a dental probe or score 0 when no plaque is present. Following this assessment, plaque score is calculated by dividing the number of plaque containing surfaces by the total number of surfaces examined.

CONTACTS AND LOCATIONS:
Overall Officials: Arif Salman, DDS, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No